CLINICAL TRIAL: NCT01854762
Title: Evaluation of the Use of Antiretroviral Regimens Containing Raltegravir for Prophylaxis of Mother-to-child-transmission of HIV Infection in Pregnant Women Presenting With Detectable Viral Load After 32 Weeks of Gestation: a Pilot Study
Brief Title: Antiretroviral Regimens Containing Raltegravir for Prophylaxis of Mother-to-child-transmission of HIV Infection
Acronym: PregnantHIV
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: IRB recommended study termination due to a significant difference between arms
Sponsor: Fundação Bahiana de Infectologia (Other)
Responsible Party: Principal Investigator, Carlos Brites, Senior Investigator, Fundação Bahiana de Infectologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PregnantHIV
Record Dates: First submitted 2013-04-22; First posted 2013-05-16 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: HIV; Pregnancy
Keywords: HIV; Treatment; Pregnancy
MeSH Terms: interventions — Raltegravir Potassium; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: Pilot randomized single-center open label clinical trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir (Experimental): Use of Raltegravir plus backbone treatment for pregnant women
  Interventions: Drug: Raltegravir
- Lopinavir/Ritonavir (Active Comparator): Use of standard PI treatment (Lopinavir/r) plus backbone treatment for pregnant women
  Interventions: Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Raltegravir — a raltegravir-based antiretroviral regimen (AZT+3TC+Raltegravir) will be administered for intervention arm patients (AZT+3TC will be administered in a fixed combination of AZT 300mg +3TC 150 mg, BID. Raltegravir will be administered in a dosis of 1 400 mg pill BID).
  Other Names: Isentress
  Arms: Raltegravir
Drug: Lopinavir/Ritonavir — The second arm (comparator)patients will use a regimen composed by AZT+3TC (same dosis/schedule of active arm)+ LPV 200mg combined with rtv 50 mg, 2 pills BID
  Other Names: Kaletra
  Arms: Lopinavir/Ritonavir

SUMMARY:
The current available antiretroviral (ARV) agents make possible a successful treatment of virtually all HIV-infected patients, even those heavily experienced subjects, with a history of previous failure to ARV drugs of different classes. However, some problems are still present, especially for specific populations, like pregnant women and infants. For these groups, most of currently available drugs are not used, because the lack of information on safety, efficacy, and pharmacokinetic/dynamic behavior of ARVs drugs. The mother to child transmission (MTCT) is still a problem in certain areas of the world, especially in resource-limited settings. In some settings, women often present to their first antenatal care visit late in the pregnancy, posing an additional problem: how to effectively treat these patients to assure they will have an undetectable viral load at the moment of delivering? Depending on the plasma viremia magnitude, and viral susceptibility it can take 6 or more weeks to reduce the viral load to less than the desired 1,000 copies of HIV-1 RNA / ml of plasma. To achieve this goal, it would be necessary the use of a potent, very efficacious ARV regimen that could provide such viral decay in a very short period. Raltegravir (RAL), the first HIV-1 integrase inhibitor, is a potent and safe ARV drug. The available evidence suggest it has no genotoxic potential, and promotes a rapid decline in HIV-1 plasma viremia. In addition, RAL is highly active against viral strains presenting different degree of resistance to other ARV drugs. Thus, RAL could be an ideal candidate to be used for prevention of MTCT for women with detectable viral load, presenting late in the course of pregnancy. Another attractive point is to consider that, due to the similarity between the integrase enzyme of HIV-1 and Human T-cell lymphotropic virus type-1 (HTLV-1); RAL could be active against HTLV-1, blocking its replication. If our hypothesis is correct, the use f RAL-containing ARV regimens would reduce the MTCT of both agents. This study has the objective of evaluating the efficacy of RAL containing ARV regimens in reducing the HIV-1 RNA plasma viral load below 50 copies/ml, at the end of pregnancy, for late-presenters pregnant women and to compare the frequency of adverse events for women using RAL-based ARV regimens and comparators, and for their babies.

DETAILED DESCRIPTION:
A total of 44 late-presenters (gestational age >28 weeks), HIV-infected pregnant women will be randomly assigned to receive an antiretroviral regimen based on Zidovudine (AZT)+Lamivudine (3TC)+Raltegravir or AZT+3TC+Lopinavir/r (LPV/r). They will be followed up to the delivery, and plasma viral load will be measured. The rate of HIV mother-to-child-transmission will be compared between groups. The newborns will be followed up to 6 months, to register any adverse event during this period of time.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with confirmed HIV-1 infection (positive Western blot or plasma HIV-1 RNA >1,000 copies/ml)
* Gestational age higher than 28 weeks
* Age equal or higher than 15 years
* HIV-1 plasma viral load ≥ 1,000 copies of HIV-1 RNA/ml

Exclusion Criteria:

* Age lower than 15 years
* Undetectable plasma viral load at screening
* Previous use of RAL

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Brites, MD, PhD, Principal Investigator — Fundação Bahiana de Infectologia
Locations (1):
- Fundação Bahiana de Infectologia/SEI, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data regarding the protocol will be made freely available at the website of Fundação Bahiana de Infectologia.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: September/1st/2017
Access Criteria: open access
URL: http://www.fbai.com.br

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir: Patients in raltegravir group received the standard dose of one 400 mg tablet twice a day, in combination with zidovudine 300 mg plus lamivudine 150 mg, in a co-formulated pill, twice a day.
- Lopinavir/Ritonavir: Participants in lopinavir/ritonavir group received two tablets containing lopinavir 200 mg plus ritonavir 100 mg twice a day, plus one zidovudine 300 mg plus lamivudine 150 mg co-formulated pill, twice a day.
Period: Overall Study
Arm/Group | Raltegravir | Lopinavir/Ritonavir
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Antiretroviral drugs-naïve, Pregnant women infected by HIV-1, with age equal or higher than18 years were eligible
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir | Lopinavir/Ritonavir | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 26.7 [18.8 to 36.7] | 26.7 [18.2 to 32.9] | 26.7 [18.2 to 36.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 0 | 2 | 2
  Black/mixed | 17 | 14 | 31
Region of Enrollment [Number; unit: participants]
  Brazil | 17 | 16 | 33
Mean Plasma HIV-1 Viral load [Median (Inter-Quartile Range); unit: copies/mL] | 12859 [5644 to 23165] | 21143 [3745 to 42750] | 15309 [4087 to 36740]
Mean CD4 count [Mean (Full Range); unit: cells/mL] | 497 [92 to 1451] | 532 [212 to 961] | 509 [92 to 1451]
Mean haemoglobin [Mean (Full Range); unit: g/dL] | 10.7 [9.2 to 13.5] | 10.7 [9.0 to 14.0] | 10.7 [9.0 to 14.0]
Gestational age [Mean (Full Range); unit: weeks] | 32.7 [28.4 to 37.2] | 32.5 [28.3 to 37.6] | 32.5 [28.3 to 37.6]

OUTCOME MEASURES:

1. Primary Outcome: HIV Viral Load at Delivery
Description: Number of participants presenting with PVL<50 copies/mL at delivery
Time Frame: 2, 4, 6 weeks and at delivery
Population: Frequency of PVL<50 copies/mL at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir | Lopinavir/Ritonavir
Number analyzed (Participants) | 17 | 16
Participants
  Frequency of VL<50 at delivery | 13 | 4
  Frequency of VL<50 at 2 weeks: number analyzed (Participants) | 17 | 15
  Frequency of VL<50 at 2 weeks | 7 | 1
  Frequency of VL<50 at 4 weeks: number analyzed (Participants) | 12 | 11
  Frequency of VL<50 at 4 weeks | 9 | 2
  Frequency of VL<50 at 6 weeks: number analyzed (Participants) | 10 | 16
  Frequency of VL<50 at 6 weeks | 10 | 4
Statistical Analysis 1: Comparison: Raltegravir vs Lopinavir/Ritonavir; Test type: Other; p < 0.01, Fisher Exact; Odds Ratio (OR) = 3.1, 95% CI 2-sided [1.3 to 7.4]; Kaplan-Meier estimates for the proportion of patients without virological failure by weeks 2, 4 and 6, and at delivery, using treatment-related discontinuation equal failure analysis

2. Secondary Outcome: Overall Adverse Events up to Delivery
Description: Frequency of clinical and laboratory abnormalities by arm
Time Frame: 2, 4, 6 weeks and at delivery
Population: Overall frequency od Adverse events
Measure: Number; unit: adverse events
Arm/Group | Raltegravir | Lopinavir/Ritonavir
Number analyzed (Participants) | 17 | 16
adverse events | 4 | 10

3. Secondary Outcome: Number of Children Infected With HIV
Description: Detectable plasma HIV-1 RNA viral load at 4 weeks after delivery
Time Frame: 4 weeks after delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir | Lopinavir/Ritonavir
Number analyzed (Participants) | 17 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: AE data were collected from baseline to delivery time (up to 8 weeks)
Description: clinical AE and laboratory AE were assessed at 2, 4 and 6 weeks and at delivery. The total number of adverse events leadinbg up to delivery, are reported
Arm/Group | Raltegravir | Lopinavir/Ritonavir
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 4/17 | 10/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=17) | Lopinavir/Ritonavir (N=16)
diarrhea (Gastrointestinal disorders) | 0 (0) | 5 (5) — diarrhea
nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) — nausea
headache (General disorders) | 0 (0) | 3 (3) — headache
miscelaneous (General disorders) | 4 (4) | 10 (13) — general complaints

LIMITATIONS AND CAVEATS:
Small sample size and current limited use of LPV/r as a first-choice drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-08-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT01854762/Prot_000.pdf
  • Statistical Analysis Plan (2011-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT01854762/SAP_001.pdf